CLINICAL TRIAL: NCT01977326
Title: The Effectiveness and Cost-effectiveness of a Task Sharing Counseling Intervention by Community Health Workers for Prenatal Depression in South Africa
Brief Title: Task Sharing Counseling Intervention by Community Health Workers for Prenatal Depression in South Africa
Acronym: AFFIRM-SA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, A/Prof Crick Lund, Professor, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5U19MH095699-02 (NIH); 1U19MH095699 (NIH)
Record Dates: First submitted 2013-10-24; First posted 2013-11-06 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Moderate Depression; Clinical Depression; Postpartum Depression
Keywords: task sharing; task shifting; prenatal depression; counselling; lay health workers
MeSH Terms: conditions — Depressive Disorder, Major; Depression, Postpartum

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- counseling intervention (Experimental): Each woman recruited into the intervention arm will undergo 6 sessions of basic counselling by lay-health workers
  Interventions: Behavioral: basic counselling by lay-health workers
- Enhanced usual care (Active Comparator): usual antenatal care with additional 3 - 4 monthly phone calls.
  Interventions: Other: Enhanced usual care

INTERVENTIONS:
Behavioral: basic counselling by lay-health workers — 6 sessions of manual based counselling by trained lay health workers
  Other Names: task sharing intervention for maternal depression
  Arms: counseling intervention
Other: Enhanced usual care — 3 monthly phone calls by trained lay health workers (without counselling)
  Arms: Enhanced usual care

SUMMARY:
The objective of this randomised controlled trial (RCT) is to determine the effectiveness and cost-effectiveness of a task sharing counseling intervention for maternal depression in South Africa(i.e. provided by non-specialist health workers)

DETAILED DESCRIPTION:
Specific Objectives:

1. To determine the effectiveness and cost-effectiveness of task sharing care to community health workers (CHWs), compared to enhanced usual care in South Africa, on both primary outcome measures (severity of prenatal maternal depression symptoms) and on a series of secondary outcome measures (functional status, health care utilization, social support and postnatal infant growth).
2. To examine factors influencing the implementation of the task sharing intervention and future scale up, by assessing feasibility, sustainability, quality, and safety, and by qualitative exploration of the experience of task sharing from the perspectives of both CHWs and patients.

ELIGIBILITY:
Inclusion Criteria:

1. Women attending antenatal clinics at the Michael Mapongwana Community Health Centre in Khayelitsha, presenting for their first booking appointment, no later than 28 weeks gestation
2. Living in Khayelitsha
3. 18 years or older
4. Screen positive for depression with a cut off of 13 or more on the EPDS
5. Able to give informed consent

Exclusion Criteria:

* Require urgent medical attention or have severe mental health problems, defined as a diagnosis of schizophrenia, bipolar mood disorder, or currently experiencing an episode of psychosis.
* Women who do not speak isiXhosa as a first language

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4205 (Actual)
Dates: Start 2013-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Hamilton depression rating Scale (HAM-D) | baseline, and change in scores at 1 month prenatally, 3 months and 12 months postnatally

SECONDARY OUTCOMES:
Edinburgh Postnatal depression scale (EPDS) | baseline and change in scores at 1 month before birth follow-up 3 months postnatal follow-up 12 months postnatal follow-up
  Screening tool to identify depressive symptoms; score of 13 or higher indicates a positive screen for depressive symptoms and woman is recruited into the study
Mini International Psychiatric Interview 2.0.0 (MINI) Major depression | baseline and change in scores at 1 month before birth follow-up 3 months postnatal follow-up 12 months postnatal follow-up
  Major Depression and Suicidality modules are used. A score of 17 or higher on the suicidality module indicates need for referral for additional treatment. These women remain in the trial.
Multidimensional Scale of Perceived Social Support (MSPSS) | baseline and change in scores at 1 month before birth follow-up 3 months postnatal follow-up 12 months postnatal follow-up
WHO Disability Assessment Schedule (WHO-DAS) 12 item version 2.0 | baseline and change in scores at 1 month before birth follow-up 3 months postnatal follow-up 12 months postnatal follow-up
Health services utilisation questionnaire | baseline and changes in scores at 1 month before birth follow-up 3 months postnatal follow-up 12 months postnatal follow-up
Cape Town Functional Assessment Instrument for Maternal Depression | baseline and changes in scores at 1 month before birth follow-up 3 months postnatal follow-up 12 months postnatal follow-up
  locally relevant functional assessment instrument developed for use with the specific target population of the trial - pregnant women and mothers of young babies living in Khayelitsha, Cape Town - the study site. This outcome measure complements the WHO-DAS 2.0
Obstetric and Infant outcome measures (head circumference, weight, height, feeding, diarrhoea, respiratory tract infections, immunisation | follow-up 3 months postnatal follow-up 12 months postnatal follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Crick Lund, PhD, Principal Investigator — University of Cape Town; Ezra Susser, PhD, Principal Investigator — Mailman School of Public Health, Columbia University; Atalay Alem, PhD, Principal Investigator — Addis Ababa University
Locations (2):
- South Africa (2):
  - Michael Mapongwana Clinic, Cape Town, Western Cape
  - Site B Clinic, Cape Town, Western Cape

REFERENCES:
- [Derived] Cleary S, Orangi S, Garman E, Tabani H, Schneider M, Lund C. Economic burden of maternal depression among women with a low income in Cape Town, South Africa. BJPsych Open. 2020 Apr 3;6(3):e36. doi: 10.1192/bjo.2020.15. PMID 32241330
- [Derived] Lund C, Schneider M, Garman EC, Davies T, Munodawafa M, Honikman S, Bhana A, Bass J, Bolton P, Dewey M, Joska J, Kagee A, Myer L, Petersen I, Prince M, Stein DJ, Tabana H, Thornicroft G, Tomlinson M, Hanlon C, Alem A, Susser E. Task-sharing of psychological treatment for antenatal depression in Khayelitsha, South Africa: Effects on antenatal and postnatal outcomes in an individual randomised controlled trial. Behav Res Ther. 2020 Jul;130:103466. doi: 10.1016/j.brat.2019.103466. Epub 2019 Oct 31. PMID 31733813
- [Derived] Munodawafa M, Lund C, Schneider M. A process evaluation exploring the lay counsellor experience of delivering a task shared psycho-social intervention for perinatal depression in Khayelitsha, South Africa. BMC Psychiatry. 2017 Jul 1;17(1):236. doi: 10.1186/s12888-017-1397-9. PMID 28666425
- [Derived] Schneider M, Baron E, Davies T, Bass J, Lund C. Making assessment locally relevant: measuring functioning for maternal depression in Khayelitsha, Cape Town. Soc Psychiatry Psychiatr Epidemiol. 2015 May;50(5):797-806. doi: 10.1007/s00127-014-1003-0. Epub 2015 Jan 8. PMID 25567235
- [Derived] Lund C, Schneider M, Davies T, Nyatsanza M, Honikman S, Bhana A, Bass J, Bolton P, Dewey M, Joska J, Kagee A, Myer L, Petersen I, Prince M, Stein DJ, Thornicroft G, Tomlinson M, Alem A, Susser E. Task sharing of a psychological intervention for maternal depression in Khayelitsha, South Africa: study protocol for a randomized controlled trial. Trials. 2014 Nov 21;15:457. doi: 10.1186/1745-6215-15-457. PMID 25416557